CLINICAL TRIAL: NCT03933787
Title: Neuropeptide Y Function in the Sympathovagal Balance During an Ergometric Test in Healthy Volunteers
Brief Title: Neuropeptide Y and Sympathovagal Balance
Acronym: NPY
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eric Grouzmann (Other)
Collaborators: grégoire wuerzner (Unknown); grégoire millet (Unknown); Nicolas Bourdillon (Unknown); Philippe Eugster (Unknown)
Responsible Party: Sponsor-Investigator, Eric Grouzmann, Head of laboratory, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2018-00569
Record Dates: First submitted 2019-04-19; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Physical Activity; Sympathetic Nervous System; Secretion; Catecholamine
Keywords: neuropeptide Y,catecholamine, exercise
MeSH Terms: conditions — Motor Activity | interventions — saxagliptin

STUDY DESIGN:
Intervention Model Description: double-blind placebo-controlled crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, investigator and care provider were not aware when the placebo or Saxagliptin was provided. The biochemical assays were performed in a random order with anonymised sample numbers. The data were analysed before revealing to which session each participant received the placebo or Sitagliptin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mannitol in a tablet (Placebo Comparator): two tablets containing mannitol in a blister: one tablet provided to each volunteer in a blister 16 hours before the trial and one tablet provided two hours before the clinical trial
  Interventions: Drug: Placebo oral capsule; Other: ergometric test in healthy volunteers
- Saxagliptin in a tablet (Active Comparator): two tablets containing each 5 mg of Saxagliptin in a blister: one tablet provided to each volunteer in a blister 16 hours before the trial and one tablet provided two hours before the clinical trial
  Interventions: Drug: Saxagliptin 5mg; Other: ergometric test in healthy volunteers

INTERVENTIONS:
Drug: Saxagliptin 5mg — Randomised study: session 1 the volunteer will receive either saxagliptin or placebo. Session 2 the volunteer will receive the placebo or saxagliptin
  Arms: Saxagliptin in a tablet
Drug: Placebo oral capsule — Randomised study: session 1 the volunteer will receive either saxagliptin or placebo. Session 2 the volunteer will receive the placebo or saxagliptin
  Arms: mannitol in a tablet
Other: ergometric test in healthy volunteers — The volunteers will undergo an ergometric test in each session

SUMMARY:
Neuropeptide Y (NPY) activates the sympathetic and vagal nervous systems through the Y1 and Y2 receptors. This double-blind placebo-controlled crossover study investigated the sympathovagal balance during three exercises on a cycloergometer in healthy volunteers treated with saxagliptin (DPP4 inhibitor).

DETAILED DESCRIPTION:
Pharmacological studies indicate that NPY has a role as a co-transmitter associated with catecholamines to maintain cardiovascular homeostasis. The development of a selective and sensitive assay of NPY1-36 (vasoconstrictor) and NPY3-36 (vasodilator) by LC-MS/MS will confirm this modulating role of NPY in sympatho vagal balance in healthy young subjects. This project should lead to a better understanding of the contribution of NPY to exercise physiology through a double-blind randomized study using a DPP4 inhibitor (Saxagliptin) used for the treatment of type 2 diabetes, blocking the formation of NPY3-36 and thus enhancing the effect of NPY1-36. The interest of this study will be to find targets other than adrenergic receptors in the regulation of sympathetic and parasympathetic systems during exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged between 18 and 30 years.
2. Non smoking
3. Practicing at least 3 hours physical activity per week
4. Absence of significant findings in the medical history and physical examination as judged by the Investigator, especially for cardiovascular, pulmonary, haematological and nervous systems
5. Ability to understand the procedures, agreement to participate and willingness to give written informed consent
6. Co-operative attitude and availability for scheduled visits over the entire study period.

Exclusion Criteria:

1. Use of any medication the week prior to study. Paracetamol is permissible before and during study as a concomitant medication but only with Investigator's permission.
2. History of major cardiovascular, pulmonary, hepatic, immunological, renal, haematological, gastrointestinal, genitourinary, neurological, or rheumatologic disorders
3. rhinosinusitis
4. Urinary tract infection
5. Hypertension defined as supine blood pressure >150/90 mmHg or recurrent hypotensive events considered as clinically relevant or documented orthostatic hypotension

Ages: 24 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Heart rate change variability assessed at the end of each exercise | 5 hours and 30 minutes
  RMSSD (Root mean square of successive RR interval differences) measurement
Heart rate change variability assessed at the end of each exercise | 5 hours and 30 minutes
  normalized low frequency (nLF) measurement

SECONDARY OUTCOMES:
NPY 1-36 secretion | 5 hours and 30 minutes
  half-life [t1/2]
NPY 1-36 secretion | 5 hours and 30 minutes
  Area under the plasma concentration versus time curve [AUC]
NPY 1-36 secretion | 5 hours and 30 minutes
  Peak Plasma Concentration [Cmax]
NPY 3-36 secretion | 5 hours and 30 minutes
  Half-life [t1/2]
NPY3-36 secretion | 5 hours and 30 minutes
  Area under the plasma concentration versus time curve [AUC]
NPY3-36 secretion | 5 hours and 30 minutes
  Peak Plasma Concentration [Cmax]
Catecholamine secretion | 5 hours and 30 minutes
  Half-life [t1/2]
Catecholamine secretion | 5 hours and 30 minutes
  Area under the plasma concentration versus time curve [AUC]
Catecholamine secretion | 5 hours and 30 minutes
  Peak Plasma Concentration [Cmax]

CONTACTS AND LOCATIONS:
Overall Officials: Eric Grouzmann, Dr, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Service de Néphrologie, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
all IPD that underlie results in a publication